CLINICAL TRIAL: NCT05600972
Title: The Efficiency of Non-FSH Versus FSH-priming in CAPA-IVM Cycles: a Randomized Clinical Trial
Brief Title: Non-FSH vs FSH-priming in Cycles With CAPA-IVM Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/22/DD-BVMD
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-03

CONDITIONS: in Vitro Maturation; FSH Priming
Keywords: in vitro maturation, FSH priming

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Embryologists are blinded to individual clinical treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-FSH priming (No Intervention): Routine CAPA-IVM treatment will be performed. The oocyte retrieval will be performed 2 days after the randomization accordingly to the current routine procedures. An ultrasound scan will be performed to exclude the development of any dominant follicle.
- FSH priming (Active Comparator): Routine CAPA-IVM treatment will be performed. Patients who are randomized into the FSH priming arm will receive two days of FSH injections of 150 IU/day. Oocyte retrieval will be scheduled at 42 hours after the last FSH injection.
  Interventions: Procedure: FSH priming

INTERVENTIONS:
Procedure: FSH priming — Patients who are randomized into the FSH priming arm will receive two days of FSH injections of 150 IU/day. Oocyte retrieval will be scheduled at 42 hours after the last FSH injection.
  Arms: FSH priming

SUMMARY:
In vitro oocyte maturation (IVM) is an assisted reproductive technology requiring minimal or no ovarian stimulation. In this technique, the immature oocytes were retrieved from follicles and subsequently cultured matured, meaning that GV oocytes reached MII in vitro (ASRM, 2021).

Currently, there is no consensus on the unique IVM protocol. However, recommended protocols that are being utilized include IVM with and without hCG (Standard IVM) and CAPA-IVM.

As mentioned previously, FSH priming before oocyte retrieval for IVM remains controversial. However, FSH is known as a hormone for the maturation of the follicles. Therefore, during oocyte maturation (IVM) cycles, FSH is used to "prime" follicular development. Generally, many studies showed a trend of a higher number of MII oocytes obtained after IVM after using FSH priming.

In animal models, Younis et al. (1994) observed a significant increase in the number of mature oocytes when performing IVM in cynomolgus monkeys (Macaca fascicularis) with a dose of 1000 IU of PMSG (pregnant mare's serum gonadotropin) in the follicular phase (Younis et al., 1994). Similarly, Wynn et al. (1998) conducted a study on mice. The results from this study revealed that a higher number of MII oocytes was observed. Still, the blastulation rate and the number of blastomeres were significantly lower than that without FSH priming. On the other hand, FSH activates meiosis resumption (Wynn et al., 1998).

In addition, an RCT of 28 patients comparing three days of 150 IU of FSH before the IVM aspiration group with the control group also showed an improvement in implantation rates in IVM cycles with FSH priming (Mikkelsen et al., 2001). The studies mentioned above both used the non-hCG IVM protocol. Other studies by Shalom-Paz et al. (2011) and Choavaratana et al. (2015) showed superiority in the number of MII oocytes.

There has been no data on the impact of not using FSH priming in CAPA-IVM cycles. Therefore, this RCT will investigate the efficacy of CAPA-IVM with and without FSH priming.

DETAILED DESCRIPTION:
3.1. Screening for eligibility and randomization

* This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Viet Nam.
* Women who are potentially eligible will be provided information about the trial at the time of IVM treatment indication.
* Screening for eligibility will be performed on the day of the first visit when the IVM treatment is indicated.
* Patients will be provided information related to the study together with the informed consent documents. Signed informed consent forms will be obtained by the investigators from all women before the enrolment.
* All patients selected for this study will undergo a 7-day COCPs administration to induce menstruation before entering both arms.
* Women will be randomized (1:1) to either non-FSH or FSH priming:

3.2 Oocytes retrieval The oocyte retrieval will be performed four days after the randomization, accordingly to the current routine procedures.

* An ultrasound scan will be performed to exclude the development of any dominant follicle.
* Patients randomized into the FSH priming arm will receive two days of FSH injections at 150 IU/day.
* Oocyte retrieval will be scheduled 42 hours after the last FSH injection.
* In the non-FSH arm, the COC will be retrieved on the same retrieval day as the FSH-treated arm.
* All the punctured follicular cohorts will be monitored carefully by ultrasound on the day before and on OPU day.

3.3 CAPA and Maturation culture: CAPA and Maturation culture will be performed routinely following current laboratory protocols.

* ICSI will be used for the fertilization of mature oocytes.
* The freeze-only will be performed, and all good embryos will be frozen on day 5 for subsequent embryo transfer.

3.4 Frozen embryo transfer After oocyte retrieval, a blister of oral contraceptive pills will be indicated to induce the bleeding.

Endometrial preparation with hormonal replacement therapy will be performed. In the following cycle, the endometrium will be prepared using oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day starting from the second or third day of the menstrual cycle. The endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Cyclogest®; Actavis) 800 mg/day will be started when endometrial thickness reached 7 mm or more. Elective single embryo transfer with a blastocyst will be performed. Embryos will be thawed on the day of embryo transfer, five days after the start of progesterone. Two hours after thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. Embryos will be transferred into the uterine cavity.

3.5 Pregnancy test and ultrasound to confirm fetal viability: A pregnancy test will be performed by measuring the blood beta-hCG level two weeks after embryo transfer. If the pregnancy test is positive (≥25mIU/mL), the patient is indicated to use exogenous estrogen (transdermal or oral) and progesterone until at least 12 weeks of gestation. A pregnancy ultrasound will be performed three weeks after the positive pregnancy test equal to 7 weeks of gestational age.

3.6 Obstetric and neonatal outcomes: All data relating to the delivery process and neonatal care will be recorded by the data management system of IVFMD.

ELIGIBILITY:
Inclusion Criteria:

* Aging from 18 to 37
* Diagnosed with PCOS followed by Rotterdam criteria
* Having an indication for CAPA-IVM treatment
* Agree to have all embryos frozen on day 5/6.
* Agree to have one blastocyst (if of good quality defined as 3BB or above) or up to two blastocysts (if no good quality are available) transferred in a subsequent frozen transfer
* Having ≤ 2 IVM/IVF attempts

Exclusion Criteria:

* A previous ovarian stimulation (for OI or IVF) within the previous three months
* Cycles with oocytes donation
* Uterine or ovarian abnormalities
* Previous evidence of a very low oocyte maturation without suspicion of FSH /LH receptor defect
* Cycles with sperms retrieved after PESA/TESE/microTESE

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Number of matured oocytes after CAPA-IVM cultured | 2 day after oocyte retrieval
  Number of oocytes at MII stage after CAPA-IVM cultured

SECONDARY OUTCOMES:
Positive pregnancy test rate | 2 weeks after embryo transfer
  A positive pregnancy test is defined as a serum human chorionic gonadotropin level greater than 25 mIU/mL. The positive pregnancy test rate is the total positive pregnancy per the number of embryos transferred.
Implantation rate | 3 weeks after embryo transfer
  Implantation rate is defined as the number of gestational sacs per the number of embryos transferred.
Ectopic pregnancy rate | 4 weeks after embryo transfer
  Ectopic pregnancy is defined as pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Clinical pregnancy rate | 5 weeks after embryo transfer
  at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Ongoing pregnancy rate | 10 weeks after embryo transfer
  Ongoing pregnancy is defined as pregnancy with a detectable heart rate at 12 weeks' gestation or beyond. The ongoing pregnancy rate is the total ongoing pregnancy per the number of embryos transferred.
Miscarriage rate | 2-10 weeks after embryo transfer
  Miscarriage is defined as the spontaneous loss of an intra-uterine pregnancy prior to 12 completed weeks of gestational age).
Live birth rate | After delivery at 12 months after randomization
  Defined as the complete expulsion or extraction from a woman of a product of fertilisation, after 24 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 350 grams or more can be used if gestational age is unknown (twins are a single count).
Multiple pregnancy rate | 5 weeks after embryo transfer
  Multiple pregnancies are defined as the presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation).
Preterm delivery rate | At delivery at 12 months after randomization
  Preterm delivery defined as delivery at <24, <28, <32, <37 completed weeks.
Birth weight | At delivery at 12 months after randomization
  including low birth weight (defined as weight < 2500 gm at birth), very low birth weight (defined as < 1500 gm at birth), high birth weight (defined as >4000 gm at birth), and very high birth weight (defined as >4500 gm at birth).
Gestational diabetes mellitus | At 24 weeks of gestation or beyond at 12 months after randomization
  Using a 75g oral glucose tolerance test
Hypertensive disorders of pregnancy | At 20 weeks of gestation or beyond at 12 months after randomization
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Antepartum hemorrhage | After delivery at 12 months after randomization
  Including placenta previa, placenta accreta, and unexplained hemorrhage
Large for gestational age | After delivery at 12 months after randomization
  Birth weight >90th centile for gestation, based on standardized ethnicity-based charts
Small for gestational age | After delivery at 12 months after randomization
  Less than 10th centile for gestational age at delivery based on standardized ethnicity-based charts
Congenital anomaly | After delivery at 12 months after randomization
  Any major congenital anomaly will be included
Perinatal mortality | After delivery at 12 months after randomization
  The death of a fetus or infant from 24 weeks of gestation to the end of the neonatal period of 4 weeks after birth.
Admission to NICU | After delivery at 12 months after randomization
  The admittance of the newborn to NICU

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, M.D., Ph.D., Principal Investigator — IVFMD and HOPE Research Center, My Duc Hospital
Locations (1):
- IVFMD - My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong LN, Ho VNA, Le AH, Nguyen NT, Pham TD, Nguyen MHN, Le HL, Le TK, Ha AN, Le XTH, Pham HH, Tran CT, Huynh BG, Smitz JEJ, Gilchrist RB, Ho TM. Hormone-free vs. follicle-stimulating hormone-primed infertility treatment of women with polycystic ovary syndrome using biphasic in vitro maturation: a randomized controlled trial. Fertil Steril. 2025 Feb;123(2):253-261. doi: 10.1016/j.fertnstert.2024.09.010. Epub 2024 Sep 12. PMID 39260537